CLINICAL TRIAL: NCT03394976
Title: Prospective Evaluation of a Rapid Diagnostic Test to Screen for Gambiense Human African Trypanosomiasis and Diagnose Plasmodium Falciparum Malaria
Brief Title: Prospective Evaluation of an RDT to Screen for Gambiense HAT and Diagnose P. Falciparum Malaria
Status: Withdrawn | Type: Observational
Why Stopped: Funding
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Makerere University (Other); Ministry of Public Health, Democratic Republic of the Congo (Other Government)
Responsible Party: Sponsor
Other Study IDs: HAT-malaria RDT evaluation
Record Dates: First submitted 2017-12-11; First posted 2018-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Human African Trypanosomiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Participants will be enrolled passively at health centres. Passive enrolment will include patients referred to or presenting directly at the health facilities.
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
A prototype rapid diagnostic test (RDT) to simultaneously screen for gambiense human African trypanosomiasis (HAT) and diagnose P. falciparum malaria (the "HAT/malaria combo") has recently been developed. The performance of this prototype has been evaluated in a retrospective study that showed that its diagnostic performance for HAT and malaria was equivalent to the performance of the SD BIOLINE HAT 2.0 and the SD BIOLINE Malaria Ag P.f tests, respectively.

The purpose of this study is to prospectively evaluate the performance of the test in settings where P. falciparum malaria is endemic, and which are either endemic or non-endemic for HAT. This will enable the assessment of the suitability of the HAT/malaria combo RDT as a diagnostic test for malaria, and a screening test for HAT in pre-elimination and post-elimination contexts, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 6 years
* Provision of signed informed consent. For children (under the age of 18) provision of signed informed consent by a parent or legal guardian and an age appropriate assent.

Exclusion Criteria:

* Severe anaemia preventing collection of a sample of venous blood
* Severe medical condition preventing informed consent and trial participation (e.g. coma, cognitive impairment, etc.)
* For HAT true negatives only: history of previous HAT infection

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be enrolled passively at health centres. Passive enrolment will include patients referred to or presenting directly at the health facilities.
  The study will focus on passive screening, which is the intended use of the test.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
specificity of the HAT/malaria combo test for gambiense HAT in passive screening | Enrolment
specificity of the SD BIOLINE HAT 2.0 test for gambiense HAT in passive screening | Enrolment
sensitivity of the HAT/malaria combo test for P. falciparum malaria in passive screening | Enrolment
sensitivity of the SD BIOLINE Malaria Ag P.f test for P. falciparum malaria in passive screening | Enrolment
specificity of the HAT/malaria combo test for P. falciparum malaria in passive screening | Enrolment
specificity of the SD BIOLINE Malaria Ag P.f test for P. falciparum malaria in passive screening | Enrolment

SECONDARY OUTCOMES:
specificity of the HAT/malaria combo test for gambiense HAT in passive screening in a population living in a setting where HAT is endemic | Enrolment
specificity of the SD BIOLINE HAT 2.0 test for gambiense HAT in passive screening in a population living in a setting where HAT is endemic | Enrolment
specificity of the HAT/malaria combo test for gambiense HAT in passive screening in a population living in a setting where HAT and animal trypanosomiasis are not endemic | Enrolment
specificity of the SD BIOLINE HAT 2.0 test for gambiense HAT in passive screening in a population living in a setting where HAT and animal trypanosomiasis are not endemic | Enrolment

IPD SHARING:
Plan to Share IPD: Undecided